CLINICAL TRIAL: NCT00667615
Title: A Multi-Center Phase I/II Trial of Vorinostat in Combination With Cyclophosphamide, Etoposide, Prednisone and Rituximab for Elderly Patients With Relapsed Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Trial of Vorinostat in Combination With Cyclophosphamide, Etoposide, Prednisone and Rituximab for Elderly Patients With Relapsed Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Northwestern University (Other); Endeavor Health (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-045
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2017-11-07 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-02

CONDITIONS: Hodgkin's Disease; Lymphoma
Keywords: vorinostat; rituximab; cyclophosphamide; etoposide; prednisone; Quality of life; 08-045
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Rituximab; Cyclophosphamide; Etoposide; Prednisone; Vorinostat; pegfilgrastim; Filgrastim

ARMS (1):
- 1 (Experimental): vorinostat in combination with cyclophosphamide, etoposide,prednisone and rituximab,peg-filgrastim or filgrastim
  Interventions: Drug: rituximab, cyclophosphamide, etoposide, prednisone, vorinostat and QOL questionnaire, peg-filgrastim or filgrastim

INTERVENTIONS:
Drug: rituximab, cyclophosphamide, etoposide, prednisone, vorinostat and QOL questionnaire, peg-filgrastim or filgrastim — Patients will be treated with 6 cycles of rituximab, cyclophosphamide, etoposide, prednisone and vorinostat every 4 weeks. Quality of life determinations will be obtained at the beginning of each cycle of chemotherapy and at each visit during the first year of followup.

SUMMARY:
The purpose of this study is to replace a drug with many side effects, procarbazine, with a new novel drug, vorinostat, in a drug combination for the treatment of patients with diffuse large B-cell lymphoma. Vorinostat is the first of a new type of chemotherapy drug, known as a histone deacetylase inhibitor, to be approved by the Food and Drug Administration. It is approved for the treatment of certain lymphomas of the skin. It alters the cancer cell pathway by preventing cancer cells from reproducing. Vorinostat will be added to a combination of four other effective chemotherapy drugs that have been used for many years for the treatment of diffuse large B-cell lymphoma: rituximab, cyclophosphamide, etoposide and prednisone. The doses of vorinostat will be increased or decreased depending on the side effects that occur in each of the first few patients in the trial to find the safest dose with the least side effects. This is termed the phase I part of the clinical trial. Once the best dose of vorinostat is found, the rest of the patients in the clinical trial will be treated with this dose. This is termed the phase II part of the trial. The object of the trial is to find out what effects, good and/or bad, the combination of vorinostat, rituximab, cyclophosphamide, etoposide and prednisone will have on you and your lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* MSKCC or Weill Cornell biopsy confirmation of relapsed/refractory diffuse large B-cell lymphoma.Patients with large cell transformation of a low-grade B-cell lymphoma will be eligible.
* One or two prior chemotherapy regimens not including autologous stem cell transplantation.
* Age ≥ 60 years.
* Not a candidate for autologous stem cell transplantation.
* Patient must have performance status of ≤2 on the ECOG Performance Scale.
* Measurable disease
* Adequate organ and bone marrow function: ANC ≥ 1000/mm3, platelet count ≥ 50,000/mm3, total bilirubin ≤ 1.5 ULN (with exception of Gilbert's disease), AST/ALT ≤ 2.5 ULN, creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 50 ml/min, potassium and magnesium within normal limits.
* Male patients agree to use an adequate method of contraception for the duration of the study.
* Patient is available for periodic blood sampling, study related assessments, and management at the treating institution for the duration of the study.

Exclusion Criteria:

* Patient who has had chemotherapy, radiotherapy, or biological therapy [including growth factors], within 30 days (42 days for nitrosoureas or mitomycin C) prior to initial dosing with study drug(s) or who has not recovered from adverse events due to agents administered more than 30 days earlier. Patients on a stable dose of steroids for at least 4 weeks prior to onset of study therapy may be included.
* Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of initial dosing with study drug(s).
* Patient had prior treatment with an HDAC inhibitor (e.g., romidespin (Depsipeptide),NSC-630176, MS 275, LAQ-824, belinostat (PXD-101), LBH589, MGCD0103,CRA024781, etc). Patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study. Patients who have received such compounds for other indications, e.g. valproic acid for epilepsy, may enroll after a 30-day washout period.
* Patients with active CNS lymphoma and/or lymphomatous meningitis are excluded. However, patients with a history of CNS lymphoma and/or lymphomatous meningitis who have been stable without evidence of CNS and/or leptomeningeal recurrence would be eligible. They must be off steroids or on a stable dose of steroids.
* Patient with a primary central nervous system lymphoma.
* Patient has known hypersensitivity to the components of study drug or its analogs.
* Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs, substance abuse or had a recent history (within the last year) of drug or alcohol abuse.
* Patient is expecting to father children within the projected duration of the study.
* Patient has uncontrolled intercurrent illness or circumstances that could limit compliance with the study, including, but not limited to the following: active infection, acute or chronic graft versus host disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric conditions.
* Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study or is not in the best interest of the patient to participate.
* Patient has a history of a gastrointestinal surgery or other procedures that might, in the opinion of the investigator, interfere with the absorption or swallowing of the study drugs.
* Patient with a "currently active" second malignancy, other than non-melanoma skin cancer and carcinoma in situ of the cervix, should not be enrolled. Patients are not considered to have a "currently active" malignancy if they have completed therapy for a prior malignancy, are disease free from prior malignancies for >5 years or are considered by their physician to be at less than 30% risk of relapse.
* Patient is HIV +.
* Patient has active hepatitis B or C.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Straus, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center @ BaskingRidge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center @ Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Relapsed or Refractory Diffuse Large B-cell Lymphoma: Patients will be treated with 6 cycles of rituximab, cyclophosphamide, etoposide, prednisone and vorinostat every 4 weeks.
Period: Overall Study
Arm/Group | Relapsed or Refractory Diffuse Large B-cell Lymphoma
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Relapsed or Refractory Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 76 [69 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Vorinostat Given Orally for 10 Days in Combination With Cyclophosphamide, Etoposide, Prednisone and Rituximab for Elderly Patients With Relapsed Diffuse Large B-cell Lymphoma
Description: Maximum Tolerated Dose (MTD) of Vorinostat reflects the highest dose of Ridaforolimus and Vorinostat that did not cause a new Grade 2 toxicity in >= 50% of participants
Time Frame: through study completion, an average of 1 year
Measure: Number; unit: mg/m2
Arm/Group | Relapsed or Refractory Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 30
mg/m2 | 300

2. Secondary Outcome: Complete Response Rate to Rituximab and a Combination of Vorinostat With Cyclophosphamide, Etoposide, and Prednisone in Elderly Pts With Relapsed Diffuse Large B-cell Lymphoma Who Aren't Candidates for Autologous Stem Cell Transplantation.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.", or similar definition that is accurate and appropriate.
Time Frame: through study completion, an average of 1 year
Measure: Number; unit: percentage of participants with CR
Arm/Group | Relapsed or Refractory Diffuse Large B-cell Lymphoma
Number analyzed (Participants) | 30
percentage of participants with CR | 32

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Relapsed or Refractory Diffuse Large B-cell Lymphoma
All-Cause Mortality (participants affected / at risk) | 25/30
Serious Adverse Events (participants affected / at risk) | 19/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relapsed or Refractory Diffuse Large B-cell Lymphoma (N=30)
Atrial fibrillation (Cardiac disorders) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Cardiac Arrhythmia, other (Cardiac disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Creatinine (Investigations) | 1
Death NOS (General disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 4
Febrile Neutropenia (Blood and lymphatic system disorders) | 6
Fever (General disorders) | 2
Hemoglobin (Investigations) | 5
Hemorrhage, Upper GI NOS (Gastrointestinal disorders) | 1
Hemorrhage (Blood and lymphatic system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infection - lung (pneumonia) (Infections and infestations) | 2
Infection - other (Infections and infestations) | 1
White blood cell (Investigations) | 4
Memory impairment (Nervous system disorders) | 1
Mucositis (func/sympt)- Stomach (Gastrointestinal disorders) | 1
Neurology - other (Nervous system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Platelets (Investigations) | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 2
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relapsed or Refractory Diffuse Large B-cell Lymphoma (N=30)
Fatigue (General disorders) | 13
Hemoglobin (Blood and lymphatic system disorders) | 13
White blood cells (Investigations) | 13
Platelets (Investigations) | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Lymphocytes (Investigations) | 11
Hyperglycemia (Metabolism and nutrition disorders) | 10
Neutrophils (Investigations) | 9
AST (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 7
ALT (Investigations) | 6
Constipation (Gastrointestinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
INR (Investigations) | 6
Nausea (Gastrointestinal disorders) | 6
Constitutional Symptoms, other (General disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Pain (General disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Alkaline phosphatase (Investigations) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 4
Hemorrhage (General disorders) | 4
Infection, other (Infections and infestations) | 4
Insomnia (Psychiatric disorders) | 4
Pain - throat (Gastrointestinal disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 4
Dysarthria (Nervous system disorders) | 4
Hyperbilirubinemia (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Edema - limb (General disorders) | 3
Fever (General disorders) | 3
Gastrointestinal, other (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Urinary frequency (Renal and urinary disorders) | 3
Vomiting (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-12-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT00667615/Prot_SAP_000.pdf